CLINICAL TRIAL: NCT01845337
Title: Toxicity OF Fluoropyrimidines: A Comparative Study of the Cardiotoxicity of capEcitabine and tEysuno
Brief Title: Study to Compare Cardiovascular Side Effects of Teysuno Versus Capecitabine
Acronym: TOFFEE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-005282-12
Record Dates: First submitted 2013-04-29; First posted 2013-05-03 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Gastrointestinal Cancer; Cancer of Unknown Primary Site; Pancreatic Cancer; Bile Duct Neoplasms
MeSH Terms: conditions — Gastrointestinal Neoplasms; Neoplasms, Unknown Primary; Pancreatic Neoplasms; Bile Duct Neoplasms | interventions — tegafur-gimeracil-oteracil; Capecitabine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Capecitabine single agent (Active Comparator): Capecitabine 1250 mg/m2 twice daily, days 1-14 every 21 days
  Interventions: Drug: Capecitabine
- Capecitabine /Oxaliplatin (Active Comparator): Capecitabine 1000 mg/m2 twice daily, days 1-14 every 21 days (in frail or elderly patients, a CAP dose of 750 mg/m2 BD should be considered). Oxaliplatin will be given as an iv infusion at a dose of 130 mg/m2 over 2-6 hours on day 1.
  Interventions: Drug: Capecitabine
- Teysuno single agent (Active Comparator): Teysuno will be administered at a dose of 30 mg/m2 twice daily, for 14 days, with a subsequent 7-day rest period. Patients will be assigned a dose on the basis of body surface area (BSA) and will receive one of the following doses twice daily: 40mg (BSA < 1.5 m2), 45 mg (BSA 1. 5 to < 1.7 m2), 55mg (BSA 1.7 - 1.9 m2),
  Interventions: Drug: Teysuno
- Teysuno/ Oxaliplatin (Active Comparator): Teysuno will be administered orally at a dose of 25mg/m2 twice daily, days 1-14 every 21 days Patients will be assigned a dose on the basis of body surface area (BSA) and will receive one of the following doses twice daily: 35mg (BSA < 1.5 m2), 40mg (BSA 1.5 to < 1.7 m2), 45mg (BSA 1.7 - 1.9 m2), 50mg (BSA >1.9 m2). Oxaliplatin will be given as an iv infusion at a dose of 130 mg/m2 over 2-6 hours on day 1.
  Interventions: Drug: Teysuno

INTERVENTIONS:
Drug: Teysuno
  Other Names: Tegafur / Gimeracil / Oteracil
  Arms: Teysuno single agent; Teysuno/ Oxaliplatin
Drug: Capecitabine
  Other Names: Xeloda tablets
  Arms: Capecitabine /Oxaliplatin; Capecitabine single agent

SUMMARY:
Capecitabine is a chemotherapy drug used to treat many types of cancer including bowel and stomach cancer. Unfortunately a side effect of this drug is that it causes heart problems including heart attacks. An alternative drug, called teysuno is used extensively in other countries instead of capecitabine and appears to have less of a bad effect on the heart whilst still killing cancer cells. This study will investigate the effect of these two drugs on the heart and blood vessels and will be the first of its kind in humans.

DETAILED DESCRIPTION:
Fluoropyrimidines (FPs) are widely used chemotherapy agents for the management of patients with colorectal, breast, upper gastrointestinal, head and neck cancers. Capecitabine is an oral prodrug of 5-fluorouracil (5FU) which is used extensively in the UK but is associated with clinically overt cardiotoxicity in up to 9% of patients. Cardiotoxicity occurs more commonly in patients with cardiovascular disease and manifests as chest pain, myocardial infarction, congestive heart failure, or sudden death with a mortality as high as 30%. In a study of continuous ECG Holter monitoring in patients receiving 5FU infusion, the majority (68%) of patients had ischaemic ECG changes and 2 patients died suddenly. We conducted a national survey of UK oncologists and 60% felt that 5FU/capecitabine cardiotoxicity was a significant problem in their clinical practice.

Hypotheses for this toxicity include ischaemia secondary to coronary artery spasm, direct endothelial cell toxicity, myocardial toxicity and interactions with the coagulation system. Studies implicate a catabolite of 5FU, in particular fluoro-alanine (FBAL). FBAL is further metabolized to fluoroacetate (FAC), a cardiac toxin that inhibits mitochondrial aconitase, resulting in cell death.

Teysuno is an oral fluoropyrimidine that has recently obtained a European licence. It is a combination of tegafur (5-FU prodrug), gimeracil (dihydropyrimidine dehydrogenase (DPD) inhibitor) and oteracil (phosphorylation inhibitor). There have been no reports of cardiac toxicity with teysuno. The incorporation of a DPD inhibitor should reduce FBAL concentrations which may prevent FP cardiotoxicity. However, this remains to be established.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at least 18 years or over with no upper age limit.
* Confirmed advanced or metastatic oesophageal, gastric, gastro-oesophageal, small bowel, colorectal, hepatobiliary or pancreatic cancer or cancer of unknown primary.
* Suitable for treatment with fluoropyrimidine, either alone or in combination with oxaliplatin.
* WHO performance status (PS) 0, 1 or 2 and considered by responsible consultant to be fit to undergo planned chemotherapy and cardiac investigations.
* Baseline laboratory tests (within 1 week prior to starting treatment):

  * Neutrophils >1.5 x109 /L and platelet count > 100 x109 /L
  * Serum bilirubin <1.5 x upper limit of normal (ULN), alkaline phosphatase <5x ULN, and serum transaminase (either AST or ALT) <3 x ULN
  * Estimated glomerular filtration rate (eGFR) >30 mL/min (Patients with eGFR 30-50 mL/min will be included but should be treated at a reduced dose (see master prescription chart).
* For women of childbearing potential; negative pregnancy test and adequate contraceptive precautions.
* Effective contraception for male patients if the risk of conception exists.
* Written informed consent for participation in the trial.

Exclusion Criteria:

* Patients who are unfit for the chemotherapy regimens in this protocol, such as:

  * Known intolerance to CAP or other FPs
  * Severe uncontrolled concurrent medical illness likely to interfere with protocol treatments
  * Poorly controlled angina or MI in previous 6 months
  * Any psychiatric or neurological condition which is felt likely to compromise the patient's ability to give informed consent or to comply with oral medication
  * Partial or complete bowel obstruction
  * Pre-existing neuropathy > grade 1 if combination therapy proposed
* Patients on therapeutic anticoagulation (warfarin or LMWH).
* Patients unable to lie flat.
* Patients unable to withstand the visits and cardiovascular investigations proposed within the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-02-05 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study will be a difference in the duration of ST deviation pre-treatment and during treatment. | Pre treatment and between day 5-7
  This will be recorded using Del Mar Reynolds Lifecard CF/Lifecard 12 recorders, which will record 12 leads over 24 hours and continuously if the storage card is changed daily. Pre-treatment control ECGs will be recorded for 24 hours. Continuous 12-lead monitoring shall be recorded for three days between day 5 and 7 of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sally Clive, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Edinburgh Cancer Centre, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) will be shared with other researchers on request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after completion of study until 5 years after archiving